CLINICAL TRIAL: NCT03342651
Title: Evaluation of the Effect of Preoperative Vitamin D Levels and Respiratory Complications of General Anesthesia
Brief Title: Preoperative Vitamin D Levels and Respiratory Complications of General Anesthesia
Acronym: VitaminD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ordu University (Other)
Responsible Party: Principal Investigator, Nilay Tas, Associate Professor, Ordu University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DVIT1
Record Dates: First submitted 2017-10-08; First posted 2017-11-17 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Vitamin D Deficiency
Keywords: Vitamin D; general anesthesia; respiratory complications
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Vitamin D; Anesthesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Observational research (Other): Vitamin D levels and respiratory complications; observational research.
  Interventions: Other: Vitamin D

INTERVENTIONS:
Other: Vitamin D — Vitamin D, general anesthesia, respiratory complications
  Other Names: Anesthesia, respiratory complications

SUMMARY:
Vitamin D deficiency is a commonly observed health problem in the world. With a role in many chronic diseases and especially lung diseases, the importance of vitamin D deficiency in anesthesia management is increased. This research aims to investigate whether there is a correlation between the respiratory complications occurring in patients under general anesthesia and preoperative vitamin D levels.

DETAILED DESCRIPTION:
This study included 95 adult cases aged from 18-65 years operated under general anesthesia. The cases had total 25-hydroxyvitamin D (25OHD) levels identified in blood samples before the operation. Patients given routine general anesthesia and postoperative monitoring procedures were assessed in terms of respiratory complications during anesthesia induction, extubation, anesthesia recovery and the first 24 hours postoperative.

This research observed that patients with low preoperative 25OHD vitamin levels encountered respiratory complications related to general anesthesia more often. Especially in the early postoperative period there is a very significant difference between complications and low 25OHD vitamin levels. Our study results show that low vitamin D levels may be a potential risk in terms of respiratory complications related to general anesthesia causing severe morbidity and mortality increase. The results lead to the consideration that optimizing vitamin D levels in the preoperative period for patients undergoing general anesthesia may aid in reducing complications.

ELIGIBILITY:
Inclusion Criteria:

- American Society of Anesthesiologists I - II risk classification, healthy adult surgery cases

Exclusion Criteria:

* Thoracic surgery, those with severe respiratory, neuromuscular or endocrine system diseases, those with difficult intubation, morbid obesity, using vitamin D supplements and those who smoked

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2016-04-01 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Relationship between Vitamin D levels and respiratory complications | Perioperative period
  Low vitamin D levels may be a potential risk in terms of respiratory complications related to general anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Nilay Taş, Assoc.Prof., Principal Investigator — Ordu University, Turkey; Tevfik Noyan, Prof., Study Chair — Ordu University, Turkey; Özgür Yağan, Assoc. Prof., Study Chair — Ordu University, Turkey; Volkan Hancı, Prof., Study Chair — Ordu University, Turkey; Ebru Çanakçı, Ass. Prof., Study Chair — Ordu University, Turkey

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hutchinson K, Healy M, Crowley V, Louw M, Rochev Y. Verification of Abbott 25-OH-vitamin D assay on the architect system. Pract Lab Med. 2017 Jan 17;7:27-35. doi: 10.1016/j.plabm.2017.01.001. eCollection 2017 Apr. PMID 28856215
- [Result] Turan A, Hesler BD, You J, Saager L, Grady M, Komatsu R, Kurz A, Sessler DI. The association of serum vitamin D concentration with serious complications after noncardiac surgery. Anesth Analg. 2014 Sep;119(3):603-612. doi: 10.1213/ANE.0000000000000096. PMID 25121616
- [Result] Holick MF, Chen TC. Vitamin D deficiency: a worldwide problem with health consequences. Am J Clin Nutr. 2008 Apr;87(4):1080S-6S. doi: 10.1093/ajcn/87.4.1080S. PMID 18400738
- [Result] Bener A, Ehlayel MS, Bener HZ, Hamid Q. The impact of Vitamin D deficiency on asthma, allergic rhinitis and wheezing in children: An emerging public health problem. J Family Community Med. 2014 Sep;21(3):154-61. doi: 10.4103/2230-8229.142967. PMID 25374465
- [Result] Columbo M, Panettieri RA Jr, Rohr AS. Asthma in the elderly: a study of the role of vitamin D. Allergy Asthma Clin Immunol. 2014 Sep 5;10(1):48. doi: 10.1186/1710-1492-10-48. eCollection 2014. PMID 25221606
- [Result] Banerjee A, Panettieri R Jr. Vitamin D modulates airway smooth muscle function in COPD. Curr Opin Pharmacol. 2012 Jun;12(3):266-74. doi: 10.1016/j.coph.2012.01.014. Epub 2012 Feb 25. PMID 22365730
- [Result] Quraishi SA, Camargo CA Jr. Vitamin D in acute stress and critical illness. Curr Opin Clin Nutr Metab Care. 2012 Nov;15(6):625-34. doi: 10.1097/MCO.0b013e328358fc2b. PMID 23075939
- [Result] Mulligan JK, Nagel W, O'Connell BP, Wentzel J, Atkinson C, Schlosser RJ. Cigarette smoke exposure is associated with vitamin D3 deficiencies in patients with chronic rhinosinusitis. J Allergy Clin Immunol. 2014 Aug;134(2):342-9. doi: 10.1016/j.jaci.2014.01.039. Epub 2014 Mar 31. PMID 24698317
- [Result] Ginde AA, Mansbach JM, Camargo CA Jr. Vitamin D, respiratory infections, and asthma. Curr Allergy Asthma Rep. 2009 Jan;9(1):81-7. doi: 10.1007/s11882-009-0012-7. PMID 19063829
- [Result] Bartley J. Vitamin D, innate immunity and upper respiratory tract infection. J Laryngol Otol. 2010 May;124(5):465-9. doi: 10.1017/S0022215109992684. Epub 2010 Jan 13. PMID 20067648